CLINICAL TRIAL: NCT06747533
Title: Impact of Diaphragmatic Breathing Coaching on Deep Inspiration Breath Hold Reproducibility and Organ Protection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1120; NCI-2024-10404 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-12-16; First posted 2024-12-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breathing, Mouth
MeSH Terms: conditions — Mouth Breathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Patient Education (Experimental): If participants are in the Standard Participants Education group, participants will receive standard of care participants education.
  Interventions: Other: CT simulation
- Breathe Radiation Protocol Coaching group (Experimental): If participants are in the Breathe Radiation Protocol Coaching group, you will have access to a video that helps guide you through a relaxed breath hold for the radiation treatment and also access to a coach for questions about the breathing process during radiation. This coaching will take place in the week before you undergo radiation planning.
  Interventions: Other: CT simulation

INTERVENTIONS:
Other: CT simulation — Given by lung function test (spirometry) and questionnaire about treatment anxiety and satisfaction.

SUMMARY:
To learn if coaching participants on diaphragmatic breathing will help participants to take larger, more reproducible breaths and feel less anxiety about their treatments.

DETAILED DESCRIPTION:
Primary Objectives The primary objective is to compare the average daily shift for participant treatment for participant who have had coaching with https://www.thebreathingclass.com/cancer-center/participant versus participant who had standard clinic teaching.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Left sided breast cancer planned for whole breast radiation or any breast cancer requiring treatment of the regional nodes
* Treatment planned at the MDACC Mays Breast Radiation Oncology clinic

Exclusion Criteria:

* Underlying lung issues that may limit ability to achieve ideal breath hold (COPD on oxygen, etc)
* Active pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women over the age of 18 with invasive breast cancer requiring radiation to the left whole breast or treatment of either the right or left breast/chestwall with comprehensive nodal irradiation will be eligible for study.
Enrollment: 40 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Mitchell, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT06747533/ICF_000.pdf